CLINICAL TRIAL: NCT06489912
Title: Etat Des Lieux de la santé Mentale Des Adolescents Suivis Par Les Dispositifs ITEP en France
Brief Title: Overview of the Mental Health of Adolescents in Therapeutci, Educational and Pedagogical Facilities in France
Acronym: PsyPreDi
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/0282/OB
Record Dates: First submitted 2024-06-28; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Mental Health Disorder
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: WAIS IV — Psychological assessement

SUMMARY:
Assess the prevalence of various psychiatric disorders in adolescents aged 12 to 16 receiving support from therapeutic, educational and pedagogical institutes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent aged 12 to 16
* In a DITEP for at least 15 days
* Minor who has been informed and has not objected to the research (according to his/her capacity)
* At least one person exercising parental authority who has read and understood the information note and has not objected to the research OR
* For a minor under guardianship: legal representative who has read and understood the information note and has not objected to the research.

Exclusion Criteria:

* Minor and/or person(s) exercising parental authority who do not understand French
* Holder of parental authority opposed to the search
* Minor opposed to search

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This is a prospective, multicentric, national cohort, including adolescents aged 12 to 16 consecutively, who have been in a French-speaking, voluntary DITEP for at least 15 days, and whose parents have given their consent.
  This choice was motivated by the fact that this is the age group most represented in Therapeutic, Educatuional and Pedagogical Institutes
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Presence of psychiatric disorders | Inclusion
  assessed according to DSM-5 by K- SADS-PL
nature of psychiatric disorders | Inclusion
  assessed according to DSM-5 by K- SADS-PL

SECONDARY OUTCOMES:
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Traumatisms
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Attachement
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Toronto Alexithymia Scale
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Empathy scale
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Impulsivity scale
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Reflective self esteem scale
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Abbreviated-diagnostic interview for borderlines
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Hostility
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Buss Durkee Hostility Inventory
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Mentoring assessed by Reflective Functioning Questionnaire
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Coping strategies assessed by Adolescent Coping Scale
Describe the psychological characteristics of adolescents aged 12 to 16 | Inclusion
  Risk behaviour assessed by COLUMBIA-SUICIDE SEVERITY RATING SCALE
cognitive abilities | Inclusion
  Raven's Matrix
Adverse exepriences | Inclusion
  Adverse Child Experiences

IPD SHARING:
Plan to Share IPD: No